CLINICAL TRIAL: NCT06442462
Title: A Randomized, Placebo-controlled, Double-blind Phase 2 Study to Assess the Efficacy, Safety, Tolerability, and Pharmacodynamics of SPG302 in Adult Participants Diagnosed With Schizophrenia
Brief Title: Study of SPG302 in Adults With Schizophrenia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Spinogenix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPG302-SCZ-201
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia
Keywords: synaptogenesis; synapse; dendritic spines
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active SPG302 to be administered to participants with Schizophrenia (Active Comparator): Participants with schizophrenia will be randomized to receive SPG302 300 mg or placebo (two capsules of 150 mg) once daily for six weeks.
  Interventions: Drug: SPG302
- Placebo comparator to be administered to participants with Schizophrenia (Placebo Comparator): Participants with schizophrenia will be randomized to receive SPG302 300 mg or placebo (two capsules of 150 mg) once daily for six weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPG302 — small synthetic molecule
  Arms: Active SPG302 to be administered to participants with Schizophrenia
Drug: Placebo — Placebo
  Arms: Placebo comparator to be administered to participants with Schizophrenia

SUMMARY:
This Phase 2 study described herein will evaluate the safety, efficacy, tolerability, and pharmacodynamics of SPG302 in adults with a primary diagnosis of schizophrenia.

DETAILED DESCRIPTION:
This Phase 2 study will evaluate the safety, efficacy, tolerability, and pharmacodynamics of SPG302 in adults with a primary diagnosis of schizophrenia. This is a randomized, placebo-controlled study of SPG302 administered once daily for six weeks.

This study will entail weekly visits to the study site for screening, study procedures, and receipt of investigational medication for use at home.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Primary diagnosis of schizophrenia
* Clinical laboratory values within normal range or < 1.5 times ULN
* Currently prescribed only one antipsychotic medication, with stable dose for at least 4 weeks
* Able and willing to provide written informed consent

Exclusion Criteria:

* Any physical or psychological condition that prohibits study completion
* Known cardiac disease
* Active or history of malignancy in the past 5 years
* History of clinically significant CNS event or diagnosis in the past 5 years.
* Receipt of investigational products within 30 days
* Blood donation within 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Symptoms Scale (PANSS Score) as determined by clinician | 6 weeks
  The PANSS is a scale to measure symptom severity of schizophrenia. Thirty symptoms of schizophrenia are evaluated by a clinician on a seven point sale, with 1 = absence of symptoms and 7 = extremely severe symptoms. This study will rate each score change by calculating the difference between baseline scale and completion of study intervention.
Electroencephalogram analysis to assess brain electrical activity | 6 weeks
  Electroencephalograms (EEG) will provide a non-invasive measurement of brain activity. This test will be used to measure specific brain responses to stimuli, including attention and decision making electrical activity and detection of unexpected changes in the auditory environment.
Change in smooth pursuit eye tracking from baseline | 6 weeks
  Participants will follow visual targets on a computer screen to assess for accuracy of following the item, and smoothness of eye movements. The visual target on the computer screen will follow several different tracking patterns and at various speeds.

SECONDARY OUTCOMES:
Safety and tolerability of SPG302 in patients with schizophrenia | 6 weeks
  Number of subjects with treatment related adverse events as assessed by analysis of adverse events including symptoms, and abnormal findings on physical examination, vital signs, ECG, and standard laboratory examination results (SAEs).
Change in Global Impressions Improvement scale as determined by clinician | 6 weeks
  Change in the Clinical Global Impression of Improvement (CGI-I) is a 3-item observer-rated scale that measures illness severity, global improvement or change, and therapeutic response. It is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients).
Change in MATRICS Consensus Cognitive Battery scale as determined by clinician | 6 weeks
  The MATRICS Consensus Cognitive Battery (MCCB) measures functioning across various cognitive domains through timed assessments. The results of each assessment are summarized for overall cognitive performance. The average score is between 40-60, and a score below 40 indicates lower overall cognitive performance.
World Health Organization Quality of Life - Abbreviated Assessment Questionnaire-brief version from baseline | 6 weeks
  This is a 26-item questionnaire which collects self-reported data on physical health, psychological health, social relationships, and environmental health. Each section is scored from 1 to 5, with higher scores indicate higher quality of life. Scores from each section are then added together for an overall score, with higher score indicating higher quality of life.
Change in Personal and Social Performance from baseline | 6 weeks
  Personal and Social Performance (PSP) evaluates overall functioning in daily life. A higher score indicates higher functioning.

CONTACTS AND LOCATIONS:
Overall Officials: David Walling, MD, Principal Investigator — CenExel
Locations (3):
- CenExel CNS, Garden Grove, California, United States
- Australia (2):
  - Box Hill Hospital - Eastern Health, Box Hill, Victoria
  - Multidisciplinary Alfred Psychiatry Research Centre (MAPrc), Melbourne, Victoria